CLINICAL TRIAL: NCT00364481
Title: Effectiveness of Tongue Exercises and Laryngopharyngeal Reflux Therapy on Upper Airway Resistance Syndrome
Brief Title: Tongue Exercises and Reflux Therapy for Upper Airway Resistance Syndrome
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Not enough subjects enrolled
Sponsor: West Side ENT (Other)
Responsible Party: Steven Park, West Side ENT
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NYEE IRB 06.06
Record Dates: First submitted 2006-08-11; First posted 2006-08-15 (Estimated); Last update posted 2012-12-20 (Estimated); Status verified 2012-12

CONDITIONS: Obstructive Sleep Apnea; Upper Airway Resistance Syndrome; Gastroesophageal Reflux
Keywords: apnea; tongue; exercises; reflux; airway; upper; fatigue
MeSH Terms: conditions — Sleep Apnea, Obstructive; Gastroesophageal Reflux; Apnea; Motor Activity; Fatigue | interventions — Omeprazole

INTERVENTIONS:
Drug: omeprazole
Behavioral: Tongue exercises

SUMMARY:
Tongue exercises are described to improved snoring and acid reflux symptoms. Acid reflux treatment has been found to improve obstructive sleep apnea to a limited degree. Upper airway resistance syndrome is caused by resistance to breathing, leading to multiple respiratory event related arousals, leading to daytime fatigue and other various physical ailments. Tongue base or retrolingual collapse is implicated in upper airway resistance syndrome. We will measure sleep quality and quality of life indices before and after treatment for subjects that undergo tongue exercises only, acid reflux treatment only, and those that undergo both treatments.

DETAILED DESCRIPTION:
Upper airway resistance syndrome (UARS) is a distinct clinical disorder characterized by repetitive arousals during sleep due to soft tissue collapse of the pharynx. It is associated with chronic daytime fatigue, insomnia, cold extremities, low blood pressure, orthostatic intolerance, headaches/migraine/TMJ, and various gastrointestinal condition. Obstructive sleep apnea (OSA) is different in that once obstruction of the pharynx occurs, there are multiple periods of complete (apnea) or incomplete cessation of breathing (hypopnea). Untreated, it has been strongly associated with daytime sleepiness, hypertension, depression, coronary artery disease, stroke, and even death. One possible mechanism of pharyngeal obstruction is that the posterior tongue is susceptible to collapse when supine during sleep, which causes further collapse of the soft palate and related structures. Acid reflux is also known to frequently coexist with UARS and OSA, possibly by increasing upper airway edema and inflammation. Treating OSA has been shown to improve reflux symptoms, and vice versa. Tongue exercises are also found to improve snoring and reflux symptoms. This study aims to validate via pre and post treatment polysomnograms, the effectiveness of tongue exercises alone, acid reflux treatment alone, or a combination of both regimens. Twenty-five patients will be randomly assigned to each of the three groups. Measurements include the percent improvement of major sleep indices within each group, as well as between groups. Quality of life variables as well as acid reflux symptom scores will be addressed as well.

ELIGIBILITY:
Inclusion Criteria:

* men and women ages 18 to 45
* supine Park tongue position 3+ or greater
* tonsil size 2 or less
* Mueller's 2+ or less
* Friedman Stage II/III
* BMI ≤ 30
* Symptoms of sleep apnea or UARS lasting for > 3 months: excessive daytime sleepiness, OR two of the following:

  * Choking or gasping during sleep
  * Recurrent awakenings from sleep
  * Unrefreshing sleep
  * Daytime fatigue
  * cold extremities
  * inability to sleep supine
  * irritable bowel syndrome / GERD / bloating
  * low blood pressure
  * orthostatic intolerance
* AHI of < 5, and RDI > 10 (polysomnogram within 1 year of entry date)

Exclusion Criteria:

* Significant nasal obstruction
* Prior pharyngeal surgery
* History of radiation to the head and neck
* Dysmorphic facies or craniofacial syndrome
* ASA class IV or V
* Major depression or unstable psychiatric disorder
* Contraindications to taking Omeprozole
* Pregnancy
* Illiteracy (unable to complete required forms)
* No phone # or mailing address, or plans to change in 3 month period
* Any further upper airway surgery within three month period

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2006-08; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Sleep quality of life indices before and after treatment for all three groups, with measurement of improvement within each group, as well as between each groups.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Y. Park, MD, Principal Investigator — New York Eye & Ear Infirmary; Omar Burschtin, MD, Study Chair — New York University; Janet M Bennett, M.Ed,CCC-SLP, Study Chair — Asheville Speech Associates